CLINICAL TRIAL: NCT05339789
Title: Long-term Surgical Treatment Outcome of Peri-implantitis Lesions
Status: Recruiting | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Medical University of Vienna (Other); Sigmund Freud PrivatUniversitat (Other); Blekinge County Council Hospital (Other)
Responsible Party: Principal Investigator, Kristina Bertl, Principal Investigator, Malmö University
Other Study IDs: 2020-01019
Record Dates: First submitted 2022-04-11; First posted 2022-04-21 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The surgical treatment outcome of patients that have been or are consecutively treated at the University of Malmö, at Blekinge hospital, and at the Dental Clinic of the Sigmund Freud University Vienna will be evaluated on an a regular base; specifically all patients treated since 2014 and those receiving treatment in the future, will be regularly assessed, max. once per year after the 1-year control from the surgical intervention for clinical and radiographic assessment of healing. Clinical peri-implant parameters (e.g., probing pocket depth) and peri-implant sulcus fluid (PISF) are collected, and a peri-apical radiographic examination is made. Further, from 200 patients treated in the future, the inflammatory peri-implant lesion will be collected and subjected to histological, microbiological, and molecular analysis. The removal of these lesions is a standard procedure and performed in all patients independent of study participation; i.e., the lesion has anyway to be removed during surgery and if the lesions are not stored, they would be thrown.

ELIGIBILITY:
Inclusion Criteria:

* All patients being treated since 2014 and continuously being treated will be called in for regular check-ups after the surgical intervention and an examination for study purpose will be performed annually.

Exclusion criteria:

- implant loss

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients being treated since 2014 and continuously being treated will be called in for regular check-ups after the surgical intervention and an examination for study purpose will be performed annually.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease resolution (Binary: yes/no) | 12 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 24 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 36 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 48 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 60 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 72 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 84 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 96 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 108 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.
Disease resolution (Binary: yes/no) | 120 months postoperative
  Disease resolution will be defined as peri-implant probing pocket depth ≤ 5 mm and no excessive bleeding and/or suppuration on probing.

CONTACTS AND LOCATIONS:
Locations (3):
- Dental Clinic, Sigmund Freud University Vienna, Vienna, Austria
- Sweden (2):
  - Blekinge hospital, Karlskrona
  - Malmö University, Malmo